CLINICAL TRIAL: NCT01108614
Title: A Randomized Community Intervention Trial on Reducing HIV Infection Among Drug Users Attending Methadone Maintenance Treatment(MMT) and Preventing Secondary Transmission From HIV Positive Clients to Their Sexual Partners in China
Brief Title: Injecting Drug Use Community Intervention Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Collaborators: Yunnan Center for Disease Control and Prevention (Other); Xinjiang Center for Disease Control and Prevention (Other); Sichuan Center for Disease Control and Prevention (Other Government); Guangxi Center for Disease Control and Prevention (Other Government); Guizhou Center for Disease Control and Prevention (Other)
Responsible Party: Professor Zunyou Wu, National Center for AIDS/STD Control and Prevention, China CDC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Drug Users Intervention; 2008ZX10001-016 (Other Grant/Funding Number: Ministry of Health, the People's Republic of China)
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-04

CONDITIONS: HIV; Hepatitis C; Syphilis; HSV-2; HIV Infections
Keywords: Methadone maintenance treatment; drug users; heroin; HIV; HCV; Syphilis; HSV-2
MeSH Terms: conditions — Hepatitis C; Syphilis; HIV Infections; Drug Misuse | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Intensive HIV psychological counseling ,Increased methadone dosage under individualized treatment principle, enhance randomized urine test, strengthen family and social support , partner notification and routine HIV testing, condom promotion, STD referral services.
  Interventions: Behavioral: Intervention
- Usual (No Intervention): Routine HIV prevention, including health education, counseling and testing, condom promotion.

INTERVENTIONS:
Behavioral: Intervention — Intensive HIV psychological counseling ,Increased methadone dosage under individualized treatment principle, enhance randomized urine test, strengthen family and social support , partner notification and routine HIV testing, condom promotion, STD referral services.
  Other Names: Comprehensive intervention group
  Arms: Intervention

SUMMARY:
The purpose of this study is to reduce the HIV/HCV incidence among the clients attending community-based methadone maintenance treatment (MMT) , and to prevent the secondary sexual transmission from HIV+ clients to their spouse and sex partners, through intensified comprehensive intervention.

DETAILED DESCRIPTION:
Even though National sentinel surveillance data show that the increase rate of HIV new infections among IDUs in China has become stabilized and slowed down, the new HIV infection is still on the rise, especially in the Yunnan, Guizhou, Guangxi, Xinjiang and Sichuan. This study attempts to further reduce the new infection among MMT clients, and particularly to prevent the transmission from HIV infected clients to their sexual partners with comprehensive intervention.

The purposes of this study are:

1. To evaluate the effectiveness of comprehensive interventions to decrease the HIV/STIs incidence among MMT clients.
2. To prevent the sexual transmission between those HIV+ clients and their spouse/partners with intensified intervention.

ELIGIBILITY:
(1) For MMT clients:

Inclusion Criteria:

* 20 years or above and have independent capacity of civil conduct.
* Those have enrolled in MMT clinics more than one month, and progressed to the phase of maintenance treatment.
* No mental and other physical diseases
* More than 6-month stay at local places and registered at the designated clinics.
* Complete Informed consent

Exclusion Criteria:

* Fail to complete Informed consent
* Temporarily transit in or out of the designated clinic.
* Those have enrolled in MMT clinics less than one month, and haven't progressed to the phase of maintenance treatment.
* With serious mental or other physical diseases

For the spouse or sex partners of MMT HIV+ clients'

Inclusion Criteria:

* 20 years or above and have independent capacity of civil conduct.
* Keep fixed sexual contact with HIV+ clients in the recent 6 month
* No mental and other physical diseases
* More than 6-month stay at local places and be able to participate the 1 year follow up.
* Complete Informed consent
* The recent HIV test is negative

Exclusion Criteria:

* Fail to complete Informed consent
* Temporarily transit in or out of the designated clinic.
* With serious mental or other physical diseases
* The recent HIV test is positive

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
HIV incidence rate | August 1,2009 to 31,Mar,2011

SECONDARY OUTCOMES:
HCV, Syphilis, HSV-2 incidence | 1,Aug.,2009 to 31,Mar,2011
MMT Retention Rate and Lapse/Relapse Rate | 1,Aug.,2009 to 31,Mar,2011
Frequency of condom uses | 1,Aug.,2009 to 31, Mar,2011
The awareness of HIV-related Information among the clients [ | 1,Aug.,2009 to 31,Mar,2011
The proportion of discordant couple/partners receiving HIV testing | 1,Aug.,2009 to 31,Dec,2010

CONTACTS AND LOCATIONS:
Overall Officials: Zunyou Wu, MD, PHD, Principal Investigator — National Center for AIDS/STD Control and Prevention, China CDC
Locations (5):
- China (5):
  - Center for Disease Control and Prevention,Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Center for Disease Control and Prevention, Guizhou Province, Guiyang, Guizhou
  - Center for Disease Control and Prevention, Sichuan Province, Chengdu, Sichuan
  - Center for Disease Control and Prevention, Xingjiang Uyghur Autonomous Region, Ürümqi, Xingjiang Uyghur Autonomous Region
  - Center for Disease Control and Prevention, Yunnan Province, Kunming, Yunnan

REFERENCES:
- [Background] Costenbader EC, Astone NM, Latkin CA. The dynamics of injection drug users' personal networks and HIV risk behaviors. Addiction. 2006 Jul;101(7):1003-13. doi: 10.1111/j.1360-0443.2006.01431.x. PMID 16771892
- [Background] Booth RE, Corsi KF, Mikulich-Gilbertson SK. Factors associated with methadone maintenance treatment retention among street-recruited injection drug users. Drug Alcohol Depend. 2004 May 10;74(2):177-85. doi: 10.1016/j.drugalcdep.2003.12.009. PMID 15099661
- [Background] Gifford E, Humphreys K. The psychological science of addiction. Addiction. 2007 Mar;102(3):352-61. doi: 10.1111/j.1360-0443.2006.01706.x. PMID 17298641
- [Background] Gyarmathy VA, Neaigus A. Marginalized and socially integrated groups of IDUs in Hungary: potential bridges of HIV infection. J Urban Health. 2005 Sep;82(3 Suppl 4):iv101-12. doi: 10.1093/jurban/jti112. PMID 16107433
- [Background] Latkin CA, Sherman S, Knowlton A. HIV prevention among drug users: outcome of a network-oriented peer outreach intervention. Health Psychol. 2003 Jul;22(4):332-9. doi: 10.1037/0278-6133.22.4.332. PMID 12940388
- [Background] Lloyd JJ, Ricketts EP, Strathdee SA, Cornelius LJ, Bishai D, Huettner S, Havens JR, Latkin C. Social contextual factors associated with entry into opiate agonist treatment among injection drug users. Am J Drug Alcohol Abuse. 2005;31(4):555-70. doi: 10.1081/ada-200068114. PMID 16320434
- [Background] Termorshuizen F, Krol A, Prins M, Geskus R, van den Brink W, van Ameijden EJ. Prediction of relapse to frequent heroin use and the role of methadone prescription: an analysis of the Amsterdam Cohort Study among drug users. Drug Alcohol Depend. 2005 Aug 1;79(2):231-40. doi: 10.1016/j.drugalcdep.2005.01.013. Epub 2005 Feb 24. PMID 16002032
- [Background] International Harm Reduction Development Program of the Open Society Institute. Saving lives by reducing harm: HIV prevention and treatment for injecting drug users. New York City, USA; 2006.
- [Background] Ball A, Beg M, Doupe A, Weiler G. World Health Organization, Evidence for Action for HIV Prevention, Treatment and Care among Injecting Drug Users. The International Journal of Drug Policy. 2005;16.
- [Background] de la Fuente L, Bravo MJ, Lew C, Barrio G, Soriano V, Royuela L. [The prevalence of human immunodeficiency virus infection and the risk behaviors in the heroin addicts of Barcelona, Madrid and Seville: an example of the advantages of centering studies on addicts and not just on intravenous users]. Med Clin (Barc). 1999 Nov 20;113(17):646-51. Spanish. PMID 10618778
- [Background] Welp EA, Lodder AC, Langendam MW, Coutinho RA, van Ameijden EJ. HIV prevalence and risk behaviour in young drug users in Amsterdam. AIDS. 2002 Jun 14;16(9):1279-84. doi: 10.1097/00002030-200206140-00011. PMID 12045494
- [Background] Garfein RS, Monterroso ER, Tong TC, Vlahov D, Des Jarlais DC, Selwyn P, Kerndt PR, Word C, Fernando MD, Ouellet LJ, Holmberg SD. Comparison of HIV infection risk behaviors among injection drug users from East and West Coast US cities. J Urban Health. 2004 Jun;81(2):260-7. doi: 10.1093/jurban/jth112. PMID 15136659
- [Background] Gilman SM, Galanter M, Dermatis H. Methadone Anonymous: A 12-Step Program for Methadone Maintained Heroin Addicts. Subst Abus. 2001 Dec;22(4):247-256. doi: 10.1080/08897070109511466. PMID 12466684
- [Background] Gogineni A, Stein MD, Friedmann PD. Social relationships and intravenous drug use among methadone maintenance patients. Drug Alcohol Depend. 2001 Sep 1;64(1):47-53. doi: 10.1016/s0376-8716(00)00230-1. PMID 11470340
- [Background] Hartel DM, Schoenbaum EE. Methadone treatment protects against HIV infection: two decades of experience in the Bronx, New York City. Public Health Rep. 1998 Jun;113 Suppl 1(Suppl 1):107-15. PMID 9722816
- [Background] Langendam MW, van Brussel GH, Coutinho RA, van Ameijden EJ. Methadone maintenance and cessation of injecting drug use: results from the Amsterdam Cohort Study. Addiction. 2000 Apr;95(4):591-600. doi: 10.1046/j.1360-0443.2000.95459110.x. PMID 10829334
- [Background] Lansky A, Abdul-Quader AS, Cribbin M, Hall T, Finlayson TJ, Garfein RS, Lin LS, Sullivan PS. Developing an HIV behavioral surveillance system for injecting drug users: the National HIV Behavioral Surveillance System. Public Health Rep. 2007;122 Suppl 1(Suppl 1):48-55. doi: 10.1177/00333549071220S108. PMID 17354527
- [Background] Brady JE, Friedman SR, Cooper HL, Flom PL, Tempalski B, Gostnell K. Estimating the prevalence of injection drug users in the U.S. and in large U.S. metropolitan areas from 1992 to 2002. J Urban Health. 2008 May;85(3):323-51. doi: 10.1007/s11524-007-9248-5. Epub 2008 Mar 15. PMID 18344002
- [Background] Des Jarlais DC, Braine N, Yi H, Turner C. Residual injection risk behavior, HIV infection, and the evaluation of syringe exchange programs. AIDS Educ Prev. 2007 Apr;19(2):111-23. doi: 10.1521/aeap.2007.19.2.111. PMID 17411414
- [Background] Des Jarlais DC, Semaan S. HIV prevention for injecting drug users: the first 25 years and counting. Psychosom Med. 2008 Jun;70(5):606-11. doi: 10.1097/PSY.0b013e3181772157. Epub 2008 Jun 2. PMID 18519886
- [Background] Gowing L, Farrell M, Bornemann R, Sullivan L, Ali R. Substitution treatment of injecting opioid users for prevention of HIV infection. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD004145. doi: 10.1002/14651858.CD004145.pub3. PMID 18425898
- [Background] Gossop M, Marsden J, Stewart D, Rolfe A. Patterns of improvement after methadone treatment: 1 year follow-up results from the National Treatment Outcome Research Study. Drug Alcohol Depend. 2000 Nov 1;60(3):275-86. doi: 10.1016/s0376-8716(00)00109-5. PMID 11053762
- [Background] King VL, Kidorf MS, Stoller KB, Brooner RK. Influence of psychiatric comorbidity on HIV risk behaviors: changes during drug abuse treatment. J Addict Dis. 2000;19(4):65-83. doi: 10.1300/J069v19n04_07. PMID 11110066
- [Background] Strang J, Marsden J, Cummins M, Farrell M, Finch E, Gossop M, Stewart D, Welch S. Randomized trial of supervised injectable versus oral methadone maintenance: report of feasibility and 6-month outcome. Addiction. 2000 Nov;95(11):1631-45. doi: 10.1046/j.1360-0443.2000.951116314.x. PMID 11219367
- [Background] Margolin A, Avants SK, Warburton LA, Hawkins KA, Shi J. A randomized clinical trial of a manual-guided risk reduction intervention for HIV-positive injection drug users. Health Psychol. 2003 Mar;22(2):223-8. PMID 12683743
- [Background] Zaric GS, Barnett PG, Brandeau ML. HIV transmission and the cost-effectiveness of methadone maintenance. Am J Public Health. 2000 Jul;90(7):1100-11. doi: 10.2105/ajph.90.7.1100. PMID 10897189
- [Background] Beckett M, Burnam A, Collins RL, Kanouse DE, Beckman R. Substance use and high-risk sex among people with HIV: a comparison across exposure groups. AIDS Behav. 2003 Jun;7(2):209-19. doi: 10.1023/a:1023906610710. PMID 14586205
- [Background] Preston KL, Umbricht A, Epstein DH. Methadone dose increase and abstinence reinforcement for treatment of continued heroin use during methadone maintenance. Arch Gen Psychiatry. 2000 Apr;57(4):395-404. doi: 10.1001/archpsyc.57.4.395. PMID 10768702
- [Background] Sees KL, Delucchi KL, Masson C, Rosen A, Clark HW, Robillard H, Banys P, Hall SM. Methadone maintenance vs 180-day psychosocially enriched detoxification for treatment of opioid dependence: a randomized controlled trial. JAMA. 2000 Mar 8;283(10):1303-10. doi: 10.1001/jama.283.10.1303. PMID 10714729